CLINICAL TRIAL: NCT04766216
Title: Overcoming Barriers to Warfarin Patient Self-management Implementation in the US Healthcare System
Brief Title: Warfarin Patient Self-management Implementation in the US Healthcare System
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Collaborators: Brigham and Women's Hospital (Other); University of Michigan (Other); VA Loma Linda Health Care System (U.S. Federal Agency); Kaiser Foundation Research Institute (Other)
Responsible Party: Principal Investigator, Daniel Witt, Professor and Chair, Department of Pharmacotherapy, University of Utah
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: IRB_00141141
Record Dates: First submitted 2021-02-16; First posted 2021-02-23 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Atrial Fibrillation; Venous Thromboembolism; Heart Valve Diseases
Keywords: Warfarin; Self-management; Implementation science; Anticoagulants
MeSH Terms: conditions — Atrial Fibrillation; Venous Thromboembolism; Heart Valve Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Warfarin Patient Self-Management (Experimental): Patients managing decisions relating to warfarin dose and next INR test based on the results of current INR test
  Interventions: Other: Patient self-management
- Historical Control (Active Comparator): Patients managed by anticoagulation providers prior to transitioning to warfarin patient self-management
  Interventions: Other: Usual care provided by anticoagulation providers

INTERVENTIONS:
Other: Patient self-management — Patient makes independent decisions regarding warfarin therapy changes using warfarin dosing tools
  Arms: Warfarin Patient Self-Management
Other: Usual care provided by anticoagulation providers — Normal care provided by anticoagulation providers
  Arms: Historical Control

SUMMARY:
In the US, patients receiving warfarin therapy are rarely allowed to engage in patient self-management (PSM) which is less burdensome, less expensive, and safer than standard clinic-directed warfarin management. The long-term objective of our application is to improve the safety of ambulatory warfarin therapy through increasing the implementation of PSM.

DETAILED DESCRIPTION:
In the US, patients receiving warfarin therapy are rarely allowed to engage in patient self-management (PSM) which is less burdensome, less expensive, and safer than standard clinician-directed warfarin management. National and international evidence-based guideline panels strongly recommend PSM over other warfarin management methods for appropriate patients because it improves INR control, cuts risk of thrombosis and death by half without increasing bleeding risk, and increases patient satisfaction and quality of life. The reasons behind PSM underutilization in US settings have not been systematically assessed and validated. We will address this knowledge gap and provide foundational information for increasing PSM utilization within the US healthcare system. Our Aim 1 will assess and validate barriers and facilitators to PSM and evaluate their applicability to the US healthcare system; Aim 2 will develop and test PSM implementation strategies in US ambulatory care sites using rapid-cycle research methodology; and Aim 3 will assess implementation (feasibility, fidelity, adoption), clinical (effectiveness, safety, equity, patient-centeredness), and end-user (satisfaction) outcomes. The long-term objective of our application is to improve the safety of ambulatory warfarin therapy through increasing the implementation of PSM. Our research proposal is guided by an implementation science logic model that incorporates well-known implementation science frameworks to support the specific aims. Qualitative data collection and analysis for Aim 1 will be organized using the Consolidated Framework for Implementation Research (CFIR) a determinant framework that identifies five domains influencing implementation: Intervention, Inner Setting, Outer Setting, Individuals, and the Implementation Process. Constructs within each domain provide guidance on factors to identify and measure as potential implementation barriers or facilitators. PSM implementation activities in Aim 2 will be guided by the Quality Implementation Framework (QIF), which identifies the critical implementation process steps and specific actions related to these steps that can be utilized to achieve quality PSM implementation. Implementation strategies will be supported by the rapid-cycle research framework developed by the AHRQ Practice Based Research Network. Implementation outcomes in Aim 3 will be structured using the well-known Reach, Efficacy, Adoption, Implementation, Maintenance (RE-AIM) framework. We will utilize a type III hybrid research design to test PSM implementation strategies while observing/gathering information on PSM-related clinical and economic outcomes.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age treated with warfarin for any indication for at least 9 months prior to enrollment
* Demonstrate the willingness and ability to test their own INR using a home INR monitoring device or have same-day access to clinic-derived INR results (e.g., via electronic medical record secure messaging)
* Willing to make independent decisions about warfarin dosing based on INR results
* Able to perform INR tests at least every 2 weeks
* Currently have and willing to maintain internet access for the duration of the study in order to complete online data collection forms
* Have an anticipated duration of warfarin therapy of at least 6 months

Exclusion Criteria:

* Goal INR range other than 2.0-3.0 or 2.5-3.5
* Known poor adherence to warfarin therapy
* Non-English speaking
* Inability or refusal to provide written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2023-03-15 (Actual); Primary Completion 2024-05-31 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
Time in therapeutic INR range (TTR) | Change from baseline at 6 months
  Percent time INR in the therapeutic range
Percent of patients transitioned to patient self-management | 6-months follow up
  Percent of patients successfully transitioned to warfarin patient self-management

SECONDARY OUTCOMES:
Episodes of major bleeding | 6-months follow up
  Episodes of bleeding meeting ISTH definition for major bleeding
Episodes of thromboembolic complications | 6-months follow
  Objectively diagnosed stroke, venous thrombosis, systemic embolism
Mental and physical health-related quality of life scores | Change from baseline at 6 months
  Mental and physical domains of quality of life as measured by the SF-12 survey
Anticoagulation therapy knowledge scores | Change from baseline at 6 months
  Scores measured by the Anticoagulation Knowledge Survey Tool
Patient satisfaction survey scores | Change from baseline at 6 months
  Patient satisfaction as measured by the Anti-Clot Treatment Scale

OTHER OUTCOMES:
Patient self-management cost effectiveness | 3-month cycles
  Cohort simulation Markov model compared to usual care

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - VA Loma Linda Healthcare System, Loma Linda, California
  - Brigham and Women's Hospital, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - University of Utah Thrombosis Center, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No